CLINICAL TRIAL: NCT02303717
Title: Improved Drug Eluting Stent for Percutaneous Coronary Intervention of the Left Main Artery in a Real World All-comers Population
Brief Title: Xience Versus Synergy in Left Main PCI
Acronym: IDEAL-LM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS National Waiting Times Centre Board (Other)
Collaborators: Boston Scientific Corporation (Industry); Venn Life Sciences (Other); Cardialysis B.V. (Industry); Diagram B.V. (Other)
Responsible Party: Principal Investigator, Prof. Keith G. Oldroyd, Consultant Cardiologist, NHS National Waiting Times Centre Board
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS Project ID162820
Record Dates: First submitted 2014-11-19; First posted 2014-12-01 (Estimated); Last update posted 2014-12-01 (Estimated); Status verified 2014-11

CONDITIONS: Coronary Artery Disease
Keywords: Left main; PCI; DES
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Xience (Active Comparator): Percutaneous coronary intervention utilising a cobalt chromium everolimus eluting stent with durable polymer (Xience) plus oral dual antiplatelet therapy (DAPT) for 12 months. DAPT will be aspirin 75-100mg daily plus either clopidogrel 75mg daily or prasugrel 5-10mg daily or ticagrelor 90mg twice daily.
  Interventions: Device: Percutaneous coronary intervention; Drug: Dual antiplatelet therapy
- Synergy (Experimental): Percutaneous coronary intervention utilising a platinum chromium everolimus eluting stent with bioresorbable polymer (Synergy) plus oral dual antiplatelet therapy (DAPT) for 4 months. DAPT will be aspirin 75-100mg daily plus either clopidogrel 75mg daily or prasugrel 5-10mg daily or ticagrelor 90mg twice daily.
  Interventions: Device: Percutaneous coronary intervention; Drug: Dual antiplatelet therapy

INTERVENTIONS:
Device: Percutaneous coronary intervention — Percutaneous coronary stent implantation
  Other Names: PCI
Drug: Dual antiplatelet therapy — Dual antiplatelet therapy with aspirin and either clopidogrel, prasugrel or ticagrelor will be recommended for 12 months duration in the Xience stent arm but only 4 months duration in the Synergy stent arm.
  Other Names: DAPT

SUMMARY:
A prospective, randomized, multicenter study in patients with an indication for coronary artery revascularisation who have been accepted for percutaneous coronary intervention (PCI) of the left main coronary artery. Patients will undergo standard PCI of the left main coronary artery and will be randomized in a 1:1 fashion to the Synergy stent or to the XIENCE stent. Dual antiplatelet therapy (DAPT) will be stopped at t=4 months in the Synergy arm whereas in the control arm DAPT will be continued for 12 months. A subgroup of 100 patients will have control angiography with Optical Coherence Tomography (OCT) at t=3 months after treatment.

DETAILED DESCRIPTION:
PCI of the left main coronary artery is a complex procedure with increased risk of both short and long-term major cardiac adverse events. With the use of coronary artery stents the outcome has significant improved and PCI of the left main is included in the European Society Cardiology guidelines [8]. However the results of first generation drug eluting stents still show significant room for improvement, as the risk of very late stent thrombosis has been shown to accrue up to 5 year follow-up. The newest generation of drug eluting stents have improved radial strength with thinner strut thickness, bioresorbable coatings for local drug delivery which are resorbed in 3 months and are applied only direct to the vessel wall. These stents have been evaluated in non-complex disease with good results. A comparison of the newest generation drug eluting stents in combination with a short duration of dual antiplatelet therapy versus current standard PCI techniques in complex PCI of left main coronary artery disease is therefore desirable.

The study stent (Synergy) is an evolution of currently used drug eluting stents and in initial trials demonstrated similar results for surrogate endpoints [4,5] On clinical endpoints no difference has been demonstrated. This results in a very small possibility of inferiority to current stents where re-intervention is the largest risk. For shortening DAPT several non-randomized studies have shown high safety with a very low risk (1%) of stent thrombosis [6]. Based on the improved properties of the study stent (biodegradable coating) the risk of early DAPT discontinuation should be minimal. For the relevant subgroup control coronary angiography with the additional use of OCT imaging can be considered a standard procedure with a very low risk of major complications (0.4%) [7] This study will investigate the short term angiographic and long term clinical outcome of after implantation of an improved drug eluting coronary artery stent (Everolimus-eluting Platinum Chromium Stent with Abluminal Bioabsorbable Polymer) with shorter post interventional dual antiplatelet therapy (DAPT) in comparison to a conventional drug eluting stent with a permanent Polymer followed by 12 months DAPT for treatment of unprotected left main coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication for coronary artery revascularisation by ESC guidelines and accepted for PCI of the left main coronary artery will be included in the study.

Main inclusion criteria:

1. Patient has an indication for coronary artery revascularisation of the left main artery in accordance with the ESC guidelines
2. Patient has been discussed with the cardiac surgeon prior to PCI procedure
3. Patient is accepted for PCI
4. Patient is at least 18 years of age.
5. The patient understands and accepts the meaning and the aims of the study and is willing to provide written informed consent
6. The patient is willing to comply with specified follow-up evaluation and can be contacted by telephone.

Exclusion Criteria:

1. Not able to receive anti-platelet treatment due to contraindications
2. Known allergy to acetylsalicylic acid, clopidogrel, prasugrel or ticagrelor
3. Cardiogenic shock
4. STEMI within the last 5 days
5. Planned surgery within 12 months after stent introduction
6. History of bleeding diathesis or active major bleedings
7. Major surgery within previous 15 days
8. Current participation in another trial which has not yet reached its primary endpoint
9. Life expectancy < 12 months
10. Hypersensitivity or contraindication to everolimus or structurally-related compounds, cobalt, chromium, nickel, tungsten, acrylic, platinum and fluoropolymers
11. Female patient with child bearing potential not taking adequate contraceptives or currently breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 818 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
MACE | 2 years
  The primary endpoint is the rate of MACE defined as death from any cause or MI or ischemia-driven target vessel revascularization (TVR) at 2 years after the procedure.

SECONDARY OUTCOMES:
All cause mortality | 2 years
  Component of the primary endpoint (MACE)
MI | 2 years
  Myocardial infarction as defined in protocol. Component of combined primary end-point (MACE)
Ischaemia driven target vessel revascularisation | 2 years
  Component of combined primary end-point (MACE)
Procedural success | 2 years
  Attainment of <30% residual stenosis of the target lesion and no in-hospital device-oriented composite endpoints (DOCE) defined as cardiac death, MI not clearly attributable to a non-treated vessel, and clinically-indicated target lesion revascularization.).
Procedural success | 3 years
  Attainment of <30% residual stenosis of the target lesion and no in-hospital device-oriented composite end-points (DOCE) as defined above at 1 month and 6 months and annually to 3 years and its individual components.
Stent thrombosis | 2 years
  Stent thrombosis according to ARC definition at all time points.
Bleeding | 2 years
  The composite of BARC 3 or 5 bleeding at 24 months according to BARC definition. The individual bleeding events (BARC 1, 2, 3, 4 and 5) according to the BARC definition

OTHER OUTCOMES:
OCT derived healing score (no units) | 3 months
  Based on 3 month OCT follow-up sub-study (n=100) OCT endpoints 3 months post-procedure (subgroup of patients) QCA parameters
Combined primary end-point in patients eligible for CABG vs patients considered inoperable | 2 years
  Secondary analysis comparing patients eligible for cardiac surgery with those deemed inoperable.
Angiographic late loss (mm) | 3 months
  Based on 3 month angiographic follow-up sub-study (n=100)